CLINICAL TRIAL: NCT00234676
Title: A Multi-Center, Double Blind, Randomized, Placebo-Controlled, Parallel Group Study for the Safety, Tolerability and Efficacy of Estrogen Replacement Therapy (Conjugated Equine Estrogens 0.625 mg Daily) in Post Menopausal Women With Parkinson's Disease
Brief Title: POETRY: Study of Estrogen Replacement Therapy in Postmenopausal Women With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Parkinson Study Group (Network)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry); Joseph and Rosalyn Newman Foundation (Unknown)
Responsible Party: Lisa Shulman, MD, Parkinson Study Group Principal Investigator
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: POETRY06032003
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2008-01-08 (Estimated); Status verified 2007-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson disease; women; postmenopause; estrogen replacement therapy; clinical trials
MeSH Terms: conditions — Parkinson Disease | interventions — Estrogens, Conjugated (USP)

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- 1 (Experimental): Premarin
  Interventions: Drug: Premarin ®

INTERVENTIONS:
Drug: Premarin ® — Premarin ® 0.625 mg per day orally

SUMMARY:
The primary objectives of the POETRY study are to assess the safety and tolerability of estrogen replacement therapy (ERT) in postmenopausal women with Parkinson's disease (PD) and to assess recruitment for a study of ERT in postmenopausal women with PD.

DETAILED DESCRIPTION:
POETRY is an 8-week study of 30 post-menopausal women with Parkinson's disease (PD) who will be enrolled at six clinical sites in the United States. The study is designed to measure the safety and tolerability of estrogen replacement therapy (ERT). The study will also measure how ERT affects thinking and behavior, movement and activities of daily living, as well as motor fluctuations and dyskinesias. Although we know there are gender differences in PD, no studies have assessed their impact on symptom management. Women with PD usually require less levodopa, are more likely to experience drug-related dyskinesia, and commonly report changes of their symptoms with menstruation, menopause and use of hormones, implying that hormonal changes may impact PD symptoms. All perimenopausal women face the decision whether or not to use estrogen replacement therapy (ERT) and for women with PD, information about estrogen's effects in PD may facilitate decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women with Parkinson's disease who experience levodopa-related motor fluctuations averaging at least 2 hours daily in the "off" state confirmed by home diaries
* Must be on a stable dose of carbidopa/levodopa, immediate or controlled release therapy, antidepressants, or anxiolytics (for the last 30 days)

Exclusion Criteria:

* Insulin dependent diabetes
* Thyroid disease

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2003-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Safety - Adverse event frequency, vital signs (change from Baseline to Month 2) | 60 days
Tolerability - Proportion of participants who complete the trial | 60 days

SECONDARY OUTCOMES:
Motor | 60 days
Cognition | 60 days
Behavior | 60 days
Serum estradiol levels - change from Baseline to Month 2 | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Shulman, MD, Principal Investigator — University of Maryland
Locations (6):
- United States (6):
  - The Parkinson's Institute, Sunnyvale, California
  - Emory University, Atlanta, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- See also: Parkinson Study Group — http://www.Parkinson-Study-Group.org